CLINICAL TRIAL: NCT07375238
Title: Effect of Daily Intake of Gazpacho on Semen Quality and Oxidative Stress in Men With Altered Semen Parameters: A Randomized Controlled Study
Brief Title: Effect of Daily Intake of Gazpacho on Semen Quality and Oxidative Stress
Acronym: G-OXSEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ginefiv (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Pablo Martí, Nurse and Dietitian-Nutritionist (Assisted Reproduction), Ginefiv
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2506-GFMAD-082-PM
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Male Infertility; Oxidative Stress; Subfertility; Oligozoospermia; Asthenozoospermia; Teratozoospermia
Keywords: Mediterranean diet; Gazpacho; sperm quality; Male infertility; Altered semen parameters; oxidative stress; OxiSperm II; Randomized trial
MeSH Terms: conditions — Infertility, Male; Infertility; Oligospermia; Asthenozoospermia; Teratozoospermia

STUDY DESIGN:
Intervention Model Description: Participants are assigned in a 1:1 ratio to either a control group following a standardized Mediterranean diet or an intervention group following the same diet with the addition of daily gazpacho intake.
Masking Description: This is an open-label study. Due to the nature of the dietary intervention, masking of participants and care providers is not feasible. Laboratory personnel performing semen analysis and oxidative stress assessments are not involved in the allocation process and are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Mediterranean Diet Alone (Control) (Active Comparator): Participants will follow a standardized Mediterranean diet for a period of 12 weeks. Adherence to the dietary recommendations will be monitored using a self-administered compliance diary and scheduled follow-up phone calls.
  Interventions: Other: Standardized Mediterranean Diet
- Gazpacho + Standardized Mediterranean Diet (Intervention) (Experimental): Participants assigned to the intervention arm will follow a standardized Mediterranean diet for 12 weeks and will additionally consume 330 mL of commercially available gazpacho once daily with a main meal. Adherence to the intervention will be monitored using a self-administered compliance diary and scheduled follow-up phone calls.
  Interventions: Other: Standardized Mediterranean Diet; Dietary Supplement: Gazpacho

INTERVENTIONS:
Other: Standardized Mediterranean Diet — Participants will follow a standardized Mediterranean diet for a period of 12 weeks. The dietary pattern emphasizes the consumption of vegetables, fruits, legumes, whole grains, olive oil as the main source of fat, moderate intake of fish and nuts, and limited intake of red and processed meats.
Dietary Supplement: Gazpacho — Participants will consume 330 mL per day of commercially available gazpacho, taken once daily with a main meal, for a period of 12 weeks. The gazpacho will be consumed as part of the daily diet in addition to a standardized Mediterranean diet.
  Arms: Gazpacho + Standardized Mediterranean Diet (Intervention)

SUMMARY:
The goal of this clinical trial is to learn whether drinking a daily serving of gazpacho can improve semen quality in men with reduced sperm quality. The study will also examine how this dietary intervention affects oxidative stress and whether it is well tolerated.

The main questions this study aims to answer are:

* Does daily consumption of gazpacho improve semen quality in men with altered semen parameters?
* Does this dietary intervention affect levels of oxidative stress in semen?
* Is daily gazpacho intake feasible and well tolerated as part of a Mediterranean diet?

Researchers will compare a Mediterranean diet plus daily gazpacho intake with a Mediterranean diet alone to determine whether adding gazpacho provides additional benefits for male reproductive health.

Participants will:

* Follow a standardized Mediterranean diet for 12 weeks
* Drink 330 mL of gazpacho every day or follow the diet without gazpacho
* Provide semen samples at the start of the study and after 12 weeks
* Complete a short diary to record adherence to the dietary intervention
* Be followed for up to 18 months to record reproductive outcomes

DETAILED DESCRIPTION:
Detailed Description

This is a single-center, prospective, randomized, open-label, parallel-group study conducted at GINEFIV (IVIRMA Madrid). Eligible participants are men aged 18-45 years with an andrological profile that includes altered semen parameters such as oligozoospermia with or without associated asthenozoospermia and/or teratozoospermia (O±A±T). Participants will be randomized in a 1:1 ratio to a control group following a standardized Mediterranean diet or an intervention group following the same diet with the addition of 330 mL per day of commercially available gazpacho.

The intervention period lasts 12 weeks. Participants in the intervention group will consume gazpacho once daily with a main meal. Two production batches of the product will be analyzed to determine lycopene, vitamin C, and vitamin E content. Adherence to the intervention will be evaluated using a self-administered compliance diary and scheduled follow-up phone calls.

Semen samples will be collected at baseline and at the end of the intervention period. Semen analysis will be performed according to World Health Organization (WHO) 2021 guidelines. Seminal oxidative stress will be assessed using the OxiSperm II test and its Research Use Only (RUO) digital application, which will not be used for clinical decision-making.

The primary objective of the study is to evaluate changes in semen quality following the intervention. Secondary objectives include the assessment of seminal oxidative stress, adherence to the dietary intervention, safety and tolerability, and reproductive outcomes collected during post-intervention follow-up.

Participants will be followed for 18 months after completion of the intervention to record reproductive outcomes. The total study duration is estimated at 54 months, including recruitment, intervention, follow-up, and data analysis periods.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 45 years
* Andrological profile including altered semen parameters such as oligozoospermia, asthenozoospermia and/or teratozoospermia (O±A±T)
* No clinical indication for sperm DNA fragmentation testing or advanced sperm selection techniques
* Willingness and ability to comply with the study protocol, including adherence to a standardized Mediterranean diet
* Signed and dated written informed consent form

Exclusion Criteria:

* Use of antioxidant supplements during the three months prior to study start.
* Active smokers or men who have stopped smoking within the last three months.
* Diagnosis of azoospermia, leucocytospermia or necrozoospermia.
* Presence of severe systemic diseases or chronic conditions that could interfere with semen quality or adherence to the study.
* Known allergy or intolerance to any ingredient of the gazpacho used in the study.
* Any medical, psychological or social condition that, in the investigator's judgement, could compromise the subject's ability to participate fully or comply with the protocol requirements.
* Simultaneous participation in another clinical study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Ejaculate Volume (mL) | Baseline to 12 weeks
  Semen volume measured according to WHO 2021 semen analysis guidelines. This outcome will be analyzed and reported as an independent measure of semen quality. No composite or aggregated semen analysis score will be calculated; each parameter will be reported separately as a standalone outcome.
Change in Sperm Concentration (million/mL) | Baseline to 12 weeks
  Sperm concentration measured according to WHO 2021 semen analysis guidelines. This outcome will be analyzed and reported as an independent measure of semen quality. No composite or aggregated semen analysis score will be calculated; each parameter will be reported separately as a standalone outcome.
Change in Total Sperm Motility (%) | Baseline to 12 weeks
  Percentage of motile spermatozoa (total motility) assessed according to WHO 2021 semen analysis guidelines. This outcome will be analyzed and reported as an independent measure of semen quality. No composite or aggregated semen analysis score will be calculated; each parameter will be reported separately as a standalone outcome.
Change in Progressive Sperm Motility (%) | Baseline to 12 weeks
  Percentage of progressively motile spermatozoa assessed according to WHO 2021 semen analysis guidelines. This outcome will be analyzed and reported as an independent measure of semen quality. No composite or aggregated semen analysis score will be calculated; each parameter will be reported separately as a standalone outcome.
Change in Normal Sperm Morphology (%) | Baseline to 12 weeks
  Percentage of spermatozoa with normal morphology assessed according to WHO 2021 criteria. This outcome will be analyzed and reported as an independent measure of semen quality. No composite or aggregated semen analysis score will be calculated; each parameter will be reported separately as a standalone outcome.

SECONDARY OUTCOMES:
Change in Seminal Oxidative Stress Signal (Color Units, CU) | Baseline to 12 weeks
  Seminal oxidative stress assessed using the OxiSperm II test based on a nitroblue tetrazolium (NBT) colorimetric reaction. The OXI II application provides a digital quantitative output expressed in Color Units (CU), ranging from 0 to 100 CU which will be reported as a continuous variable.
Adherence to Gazpacho Intake (%) | Baseline to12 weeks
  Percentage of planned gazpacho intakes completed during the 12-week intervention period, assessed using a self-administered compliance diary and scheduled follow-up phone calls.
Incidence of Treatment-Emergent Adverse Events | Baseline to 12 weeks
  Number and type of adverse events reported by participants during the 12-week dietary intervention period, assessed through participant self-report and scheduled follow-up phone calls.
Biochemical Pregnancy Rate | Up to 18 months post-intervention
  Proportion of female partners with at least one positive serum or urinary hCG test during the follow-up period, calculated as the number of participants with a biochemical pregnancy divided by the total number of participants at risk.
Clinical Pregnancy Rate | Up to 18 months post-intervention
  Proportion of female partners with an ultrasound-confirmed intrauterine pregnancy during the follow-up period, calculated as the number of participants with a clinical pregnancy divided by the total number of participants at risk.
Miscarriage Rate | Up to 18 months post-intervention
  Proportion of clinically confirmed pregnancies that result in pregnancy loss, calculated as the number of miscarriages divided by the total number of clinical pregnancies.
Live Birth Rate | Up to 18 months post-intervention
  Proportion of pregnancies resulting in a live-born infant, calculated as the number of live births divided by the total number of clinical pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Martí Pastor, RD, RND, Principal Investigator — Ginefiv Madrid (IVIRMA Group)
Locations (1):
- GINEFIV Madrid (IVIRMA Group), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with external researchers. The study involves sensitive reproductive health data, and there is no predefined plan for public data sharing. Data may be processed by authorized technical partners for analytical purposes under confidentiality agreements, in compliance with applicable data protection regulations.